CLINICAL TRIAL: NCT01921114
Title: A Randomized Prospective Multicenter Evaluation to Investigate the Incidence of Catheter Related Venous Thrombosis in Patients Undergoing Intravenous Therapy With the BioFlo™ Peripherally Inserted Central Catheter (PICC) or Bard® Dual-Lumen PowerPICC SOLO2®
Brief Title: The PROOF Study: The PICC Related Obstruction Of Flow Study
Acronym: PROOF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VA-BF400
Record Dates: First submitted 2013-08-08; First posted 2013-08-13 (Estimated); Results first posted 2019-05-17 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Patients Indicated for a PICC for Any Medical Condition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- BioFlo™ PICC (Active Comparator): BioFlo™ Peripherally Inserted Central Catheter (PICC)
  Interventions: Device: BioFlo™ Peripherally Inserted Central Catheter (PICC)
- Bard® PowerPICC SOLO2® (Active Comparator): Bard® Dual-Lumen PowerPICC SOLO2®
  Interventions: Device: Bard® Dual-Lumen PowerPICC SOLO2®

INTERVENTIONS:
Device: BioFlo™ Peripherally Inserted Central Catheter (PICC)
  Arms: BioFlo™ PICC
Device: Bard® Dual-Lumen PowerPICC SOLO2®
  Arms: Bard® PowerPICC SOLO2®

SUMMARY:
The main purpose of this study is to confirm whether the AngioDynamics BioFlo™ Peripherally Inserted Central Catheter (PICC) is associated with less formation of blood clots compared to another commercially available PICC.

DETAILED DESCRIPTION:
Purpose:

To investigate whether the BioFlo™ PICC will be associated with a reduced incidence of catheter-related venous thrombosis (including both symptomatic and asymptomatic) compared to another commercially available PICC: the Bard® PowerPICC SOLO2®

Design:

This is a randomized, multi-center clinical study. The study is designed as a two-arm prospectively controlled trial. Participants will be randomly assigned to either the study or control catheter using a 1:1 schema.

Enrollment:

Four hundred sixteen (416) patients will be enrolled at four (4) to eight (8) study sites in order to obtain 354 evaluable patients.

Study Objectives:

The primary objective of this study is to investigate the incidence of catheter-related venous thrombosis in patients receiving either the 5 Fr BioFlo™ PICC catheter or the control catheter, i.e., the 5 Fr Dual-Lumen PowerPICC SOLO2® catheter.

Secondary objectives of this study are to investigate:

* Incidence of other catheter-related complications, inclusive of catheter occlusion, catheter-related infection, technical failures, and premature catheter removals
* Incidence of catheter occlusion (independently from other catheter-related complications)

Additionally, economic outcomes with respect to medical resource utilization requirements will be compared between the two catheter groups (at US sites only).

ELIGIBILITY:
Inclusion Criteria:

1. Is indicated for a PICC based on institutional practices
2. Is ≥ 18 years of age
3. Is expected to require use of a PICC for a minimum of 10 days
4. Has normal findings on initial ultrasonography (complete Ultrasound Checklist)
5. Vein used for PICC placement must be a minimum of 5mm in diameter
6. Is able to comprehend and have signed the Informed Consent Form (ICF) to participate in the study (or has the ICF signed by the patient's legal representative)

Exclusion Criteria:

1. Anticipates or has presence of dialysis grafts or other ipsilateral intraluminal devices, including pacemakers (with the exception of peripheral IV catheters)
2. Has current or anticipated hematologic derangements, including:

   * thrombocytopenia
   * history of heparin-induced thrombocytopenia
   * coagulopathy (International Normalized Ratio 2.5 or greater)
   * established diagnosis of hypercoagulable syndrome (e.g., protein C and S deficiency, anti-phospholipid antibody or polycythemia) or requires systemic therapeutic anticoagulation (Note: The following prophylactic treatments are allowed: subcutaneous heparin or enoxaparin sodium injection, and concomitant use of platelet aggregation inhibitors, e.g., Plavix/Ticlid/aspirin)
3. Has central veno-occlusive disease
4. Has history of previous catheter-related thrombosis
5. Has arm identified for catheterization that exhibits any of the following (and the contralateral arm is also unsuitable for PICC placement based on the same criteria):

   * Current (or prior history of) venous thrombosis in all or any portion of the vein where the catheter is expected to reside
   * Conditions that impede venous return from the extremity (such as paralysis or lymphedema after mastectomy)
   * Pre-existing skin surface or subsurface infection at or near the proposed catheter insertion site
   * Anatomical distortions from surgery, injury or trauma (e.g., orthopedic conditions such as compound fractures requiring reconstructive procedures)
   * Anatomical irregularities (structural, vascular, neurological) which may compromise catheter insertion or catheter care procedures in the involved extremity (e.g., reflex sympathetic dystrophy)
6. Is pregnant or lactating
7. Has been previously enrolled in this clinical study, or is participating in another clinical study that is contraindicative to the treatment or outcomes of this investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Hahn, MD, Principal Investigator — Endeavor Health
Locations (5):
- United States (3):
  - University of Miami Hospital, Miami, Florida
  - NorthShore University HealthSystem, Evanston, Illinois
  - University of Louisville/Norton Hospital, Louisville, Kentucky
- Ottawa Hospital, Ottawa, Ontario, Canada
- Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne, Switzerland

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was prematurely terminated and the PI was blinded to study data, and therefore never had access to the data and does not have any information that might help us locate it. Additionally, AngioDynamics' IT team ran a thorough search for any data related to this study and no results were found.
Period: Overall Study
Arm/Group | BioFlo™ PICC | Bard® PowerPICC SOLO2®
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was prematurely terminated and the PI was blinded to study data, and therefore never had access to the data and does not have any information that might help us locate it. Additionally, AngioDynamics' IT team ran a thorough search for any data related to this study and no results were found.
Groups:
- Total: Total of all reporting groups
Arm/Group | BioFlo™ PICC | Bard® PowerPICC SOLO2® | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Catheter-related Venous Thrombosis as Confirmed by Diagnostic Ultrasound
Time Frame: 10 (+/-3) days and any time there is clinically suspected venous thrombosis (as per standard of care)
Population: as for baseline characteristics
Arm/Group | BioFlo™ PICC | Bard® PowerPICC SOLO2®
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Incidence of Other Catheter-related Complications
Description: Secondary objectives of this study are to investigate:
  * Incidence of other catheter-related complications, inclusive of catheter occlusion, catheter-related infection, technical failures, and premature catheter removals
  * Incidence of catheter occlusion (independently from other catheter-related complications)
Time Frame: Up to 30 days post-insertion
Population: as for baseline characteristics
Arm/Group | BioFlo™ PICC | Bard® PowerPICC SOLO2®
Number analyzed (Participants) | 0 | 0

3. Other Pre Specified Outcome: Medical Resource Utilization Data Analysis
Description: Economic outcomes with respect to medical resource utilization requirements will be compared between the two PICC groups. Only data from US sites will be used for this analysis.
Time Frame: Up to 30 days post-insertion
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: The study was prematurely terminated and the PI was blinded to study data, and therefore never had access to the data and does not have any information that might help us locate it. Additionally, AngioDynamics' IT team ran a thorough search for any data related to this study and no results were found.
Arm/Group | BioFlo™ PICC | Bard® PowerPICC SOLO2®
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was prematurely terminated and any data related to this study has been lost.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less